CLINICAL TRIAL: NCT03109405
Title: A Prospective, Single Center, Randomized, Cross-over Clinical Trial to Assess the Safety and Effectiveness of the Veinplicity Venous Access Device
Brief Title: Assess Veinplicity Venous Access Device Safety and Effectiveness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Physeon GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: 292-13-280681
Record Dates: First submitted 2016-04-21; First posted 2017-04-12 (Actual); Last update posted 2018-04-05 (Actual); Status verified 2018-04

CONDITIONS: Phlebotomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- stimulation-assisted (Experimental): All subjects received treatment (stimulation-assisted) with the Veinplicity Device per the Instructions for Use. The subject underwent standard IV cannulation using a 20 gauge cannula into the available vein immediately after completion of device stimulation. Use of a tourniquet was at the discretion of the nurse performing the IV cannulation.
  Interventions: Device: Stimulation-assisted venous access; Other: 20 guage cannula for IV, tourniquet optional
- standard IV cannulation (Other): The subject underwent standard IV cannulation using a 20 gauge cannula into the best available vein. Use of a tourniquet was at the discretion of the nurse performing the IV cannulation.
  Interventions: Other: 20 guage cannula for IV, tourniquet optional

INTERVENTIONS:
Device: Stimulation-assisted venous access — Stimulation-assisted venous access
  Other Names: Veinplicity Device
  Arms: stimulation-assisted
Other: 20 guage cannula for IV, tourniquet optional — Standard IV cannulation using 20 ga needle, and use of tourniquet at discretion of nurse performing IV cannulation

SUMMARY:
The purpose of this study was to examine the Veinplicity Device as an adjunctive IV cannulation tool in subjects with a history of difficult to access veins. The Veinplicity Device is intended to improve venous access rates in compromised patients by taking advantage of the increased circulation that results from provoked muscle stimulation. The study collected information about the device, intravenous access, user and patient perceptions for IV access, and any device or procedural complications or other adverse events. Device use was examined with patients in both a prone and upright position.

ELIGIBILITY:
Inclusion Criteria:

* Subject ≥ 18 years of age
* Subject with history of failed venous access, venipuncture, or IV cannula placement
* Subject agreed to required follow-up
* Subject provided written, informed consent

Exclusion Criteria:

* Subject currently had compromised skin on either forearm or hand
* Subject currently on any blood thinning medication other than 81mg of aspirin
* Subject had been diagnosed with peripheral neuropathy, has had a complex fracture or surgery in the forearm, or has other condition that diminishes sensation in one or both arms, hands or fingers
* Subject had a demand type pacemaker or defibrillator
* Subject is female of child-bearing potential and had a positive urine pregnancy test
* Subject had a history of seizure, convulsions or epilepsy
* Subject had a known allergy to Epsom salts
* Subject had any other condition that may affect the ability to complete study requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2015-06; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Rate of successful venous access on the first attempt. | 7 days
Rate of adverse events associated with either the treatment or the venous access site. | 7 days

SECONDARY OUTCOMES:
User Perception of IV cannulation difficulty, | 7 days
Subject Preception of IV cannulation pain | 7 days
Subject Perception of Device stimulation | 7 days
Time required to achieve successful IV cannula placement | time from initial puncture to successful IV cannulation
Number of attempts required to achieve successful IV cannula placement | over a 24 hour period
  number of punctures from initial puncture to successful IV cannulation

CONTACTS AND LOCATIONS:
Overall Officials: Leela Vrishabhendra, MD, Principal Investigator — Medpace Medical Device

IPD SHARING:
Plan to Share IPD: No